CLINICAL TRIAL: NCT03890497
Title: Assessment of Poliovirus Type 2 Immunogenicity of One and Two Dose Schedule With IPV and fIPV
Brief Title: Assessment of Poliovirus Type 2 Immunogenicity of One and Two Dose Schedule With IPV and fIPV When Administered at 9-13 Months of Age in Bangladesh
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Collaborators: World Health Organization (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PR-18016
Record Dates: First submitted 2019-03-19; First posted 2019-03-26 (Actual); Last update posted 2022-04-13 (Actual); Status verified 2022-03

CONDITIONS: Poliomyelitis
MeSH Terms: conditions — Poliomyelitis

STUDY DESIGN:
Intervention Model Description: • To assess the seroconversion to PV2 after one and two doses of fIPV and IPV when first dose is administered to children aged between 9 and 13 months with second dose administered 2 months later.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Full dose of IPV (Active Comparator): IPV first dose between 9 -13 months with second dose administered 2 months later.
  Interventions: Biological: IPV
- Fractional Dose of IPV (Active Comparator): fIPV first dose between 9 -13 months with second dose administered 2 months later
  Interventions: Biological: IPV

INTERVENTIONS:
Biological: IPV — The inactivated poliovirus vaccine (IPV) developed by Salk was the first available polio vaccine licensed in 1955 in the United States. The current formulation of IPV got licensed in 1987 and has a higher potency than the original Salk IPV. Almost 100% of children two months of age or older who receive 2-3 doses of intramuscular (IM) IPV achieve high antibody levels against the all three serotypes. IPV (.5mL) can be administered subcutaneously (SC) or IM and fractional (0.1 ml) doses of IPV are generally administered intradermally
  Other Names: fIPV

SUMMARY:
Following a recommendation on October 2017 meeting of the Strategic Advisory Group of Experts (SAGE) on Immunization; low- risk bOPV-using countries may adopt 2 dose fIPV schedule prior to global OPV cessation as it provides better seroconversion than 1 full dose IPV and in the post-cessation era, the 2 fIPV doses will provide sufficient (above 90%) seroconversion. Countries, which delayed the introduction of IPV or had a vaccine stock-out, should provide 1 full dose or 2 fIPV doses to all children who were missed as soon as supply becomes available. The IPV supply situation is expected to improve in 2018; all countries are expected to have access to IPV for their routine immunization programmes from the end of the first quarter of 2018.

While immunogenicity after one and two doses of IPV and fIPV has been estimated when administered to younger children ; the immunogenicity of IPV (or fIPV) when administered at 9 months of age or later is not known. We propose to conduct a study to assess the immunogenicity of one and two doses of fIPV and IPV when administered between 9-13 months of age.

ELIGIBILITY:
Inclusion Criteria:

1. Apparently healthy children with no obvious clinical symptom of illness
2. Parents/legal guardians of participants willing to give written informed consent and willing to comply with study protocol.
3. Free of obvious health problems (congenital abnormalities, severe malnutrition, acute or chronic diarrhea, bleeding disorder etc) as established by medical history and screening evaluation including clinical examination.
4. Resident of study area.

Exclusion Criteria:

1. Participation in another clinical trial in the 4 weeks preceding the (first) trial vaccination or planned participation in another clinical trial during the present trial period.
2. A diagnosis or suspicion of congenital or acquired immunodeficiency disorder, malignancy,
3. A diagnosis or suspicion of bleeding disorder
4. Acute or persistent diarrhoea
5. History of allergy or systemic hypersensitivity to any of the vaccine components
6. Chronic illness at a stage that could interfere with trial conduct or completion.
7. Presence of significant malnutrition
8. History of any neurological disorder or history of seizure (febrile or afebrile), or encephalopathy, encephalitis, hypotonic-hyporesponsive episode.

09. Febrile illness or acute illness on the day of inclusion

-

Ages: 9 Months to 13 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 300 (Estimated)
Dates: Start 2018-09-27 (Actual); Primary Completion 2022-09 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
Seroconversion to PV2 two months after the first fIPV or IPV dose | 2 months

CONTACTS AND LOCATIONS:
Locations (2):
- Bangladesh (2):
  - Matlab Health Research Centre, Chāndpur
  - Mirpur Study clinic, Dhaka

REFERENCES:
- [Derived] Aziz AB, Verma H, Jeyaseelan V, Yunus M, Nowrin S, Moore DD, Mainou BA, Mach O, Sutter RW, Zaman K. One Full or Two Fractional Doses of Inactivated Poliovirus Vaccine for Catch-up Vaccination in Older Infants: A Randomized Clinical Trial in Bangladesh. J Infect Dis. 2022 Oct 17;226(8):1319-1326. doi: 10.1093/infdis/jiac205. PMID 35575051